CLINICAL TRIAL: NCT01825759
Title: The Impact of Compound Danshen Dropping Pill for Coronary Heart Disease With Hypertension Patient Heart and Artery Structure and Function
Brief Title: Danshen Dropping Pill for Coronary Heart Disease Heart and Artery Structure and Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Compound danshen dropping pill for coronary heart disease with hypertension patient heart and artery structure and function, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: West China Hospital
Record Dates: First submitted 2013-03-26; First posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Heart Disease; Essential Hypertension
MeSH Terms: conditions — Coronary Disease; Essential Hypertension | interventions — danshen dripping pill

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- danshen dripping pill (Experimental): danshen dripping pill 27mg ten pills by mouth every 8 hours for one year
  Interventions: Drug: danshen dripping pill

INTERVENTIONS:
Drug: danshen dripping pill
  Other Names: compound danshen dripping pill

SUMMARY:
The Impact of Compound danshen dropping pill for coronary heart disease (CHD) heart and artery structure and function in patients with hypertension

DETAILED DESCRIPTION:
Compound danshen dropping pill for coronary heart disease (CHD) heart and artery structure and function in patients with hypertension.We can accorand the pwv ,IMT and MDA to assess the impact of heart and artery structure and function.

ELIGIBILITY:
Inclusion Criteria:coronary heart disease，primary hypertension， -

Exclusion Criteria:secondary hypertension，diabetes mellitus，chronic renal disease，cardiac insufficiency

-

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | one year

SECONDARY OUTCOMES:
ankle-brachial index | one year

OTHER OUTCOMES:
intima-media thickness,methyl-di-aide-hyde | one year

CONTACTS AND LOCATIONS:
Overall Officials: chen xi ping, master, Study Director — organizer
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- See also: ABI — http://ClinicalTrials.gov
- See also: IMT — http://ClinicalTrials.gov